CLINICAL TRIAL: NCT00868699
Title: A Randomized, 6-Week, Double-Blind, Placebo-Controlled, Fixed-Flexible Dose, Parallel-Group Study of Lurasidone for the Treatment of Bipolar I Depression
Brief Title: Lurasidone - A 6-week Study of Patients With Bipolar I Depression (Monotherapy)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1050236; EUDRACT No. 2008-007457-13
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Bipolar Depression
Keywords: Bipolar I, Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- lurasidone low arm (Experimental)
  Interventions: Drug: lurasidone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- lurasidone high arm (Experimental)
  Interventions: Drug: lurasidone

INTERVENTIONS:
Drug: lurasidone — lurasidone 20 mg/day for Days 1-2, 40 mg/day for Days 3-4, 60 mg/day for Days 5-6 and 80 mg/day on Day 7 and 80-120 mg/day
  Arms: lurasidone high arm
Drug: lurasidone — lurasidone 20 mg/day for Days 1-7
  Arms: lurasidone low arm
Drug: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
This clinical study is designed to test the hypothesis that lurasidone is effective, tolerable, and safe for the treatment of patients with bipolar I depression

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with bipolar I disorder, most resent episode depressed
* Subject must have a lifetime history of at least one bipolar manic or mixed episode

Exclusion Criteria:

* History of nonresponse to an adequate (6-week) trial of three or more antidepressants (with or without mood stabilizers) during the current episode
* Subject has been hospitalized for a manic or mixed episode within 60 days prior to randomization
* Imminent risk of suicide or injury to self, others, or property

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2009-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (55):
- United States (22):
  - Synergy Escondido,710 East Grand Ave., Escondido, California
  - Collaborative Neuroscience Network Inc.,12772 Valley View Street,Suite 3, Garden Grove, California
  - Excell Research, Inc,3998 Vista Way,Suite 100, Oceanside, California
  - University of California at Irvine Medical Center, Orange, California
  - California Neuropsychopharmacology,CNRI - Los Angeles LLC,8309 Telegraph Road, Pico Rivera, California
  - California Neuropsychopharmacology Clinical Research Institute, LLC,466 26th Street,6th Floor, San Diego, California
  - University of Colorado, Aurora, Colorado
  - Florida Clinical Research Center, LLC,3914 State Road 64 East, Bradenton, Florida
  - Florida Clinical Research Center, LLC,2300 Maitland Center Parkway,Suite 230, Maitland, Florida
  - Depression and Anxiety Disorders Research Institute, Tampa, Florida
  - Janus Center for Psychiatric Research,5601 Corporate Way,Suite 103, West Palm Beach, Florida
  - American Medical Research Inc.,1200 Harger Road Suite 415, Oak Brook, Illinois
  - Lake Charles Clinical Trials LLC,2770 3rd Avenue,Suite 340, Lake Charles, Louisiana
  - Sheppard Pratt Health System,6501 North Charles Street, Baltimore, Maryland
  - Albuquerque Neuroscience Inc., 101 Hospital Loop, NE, Suite 209, Albuquerque, New Mexico
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richard H. Weisler., M.D., P.A., & Associates,700 Spring Forest Road,Suite 125, Raleigh, North Carolina
  - Mood Disorders Program-UHCMC, Cleveland, Ohio
  - MetroHealth System, Cleveland, Ohio
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - FutureSearch Clinical Trials, LLC.,4200 Marathon Blvd.,Suite 200, Austin, Texas
- Czechia (4):
  - Medical Services Prague s.r.o., Kolejni 429-5, Prague
  - Psychiatricka ambulance, Brno - Mesto
  - BIALBI s.r.o., Psychiatricke Oddeleni, Litoměřice
  - Clintrial, s.r.o., Prague
- France (2):
  - Hopital Caremeau, Service de Psychiatrie A, Nîmes
  - Zans Ritter, Marcel, Orvault
- India (9):
  - S V Medical College, Tirupati, Andh Prad
  - Vijayawada Institute of Mental Health and Neurosciences, Psychiatry, Vijaywada, Andh Prad
  - Samvedna Hospitals, Ahmedabad, Gujarat
  - Seth K M School of P G Medicine & Research, Ahmedabad, Gujarat
  - Mental Illness Treatment Rehabilitationi Foundation, Ahmedabad, Gujarat
  - Spandana Nursing Home, Bangalore, Karna
  - Sujata Birla Hospital & Research Centre, Nashik, Mahara
  - R.K. Yadav Memorial Mental Health & De-Addiction Hospital, Jaipur, Rajasthan
  - Manobal Med. Research Centre, Lucknow, Uttar Prad
- Romania (5):
  - Spitalul Clinic de Urgenta Militar Central, Bucdresti
  - Spitalul Clinic de Psihaiatrie Prof. Dr. Alexandru Obregia, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca
  - Spitalul Clinic de Neuropsihiatrie Craiova, Craiova
  - Spitalul Clinic de Neurologie si Psihiatrie Oradea, Oradea
- Russia (3):
  - City Psychiatric Hospital #2 of St. Nikolay Chudotvorets, Saint Petersburg
  - Bekhterev Scientific Research Psychoneurological Institute, Saint Petersburg
  - Psychoneurology Dispensary #4, Saint Petersburg
- South Africa (5):
  - Cape Trial Centre, Cape Town, W. Cape
  - Paarl Medical Centre, Paarl, W. Cape
  - Clinika, Port Elizabeth, E. Cape
  - Dey Clinic, Pretoria, Gauteng
  - Vereeniging Medi-Clinic, Vereeniging, Free State
- Ukraine (5):
  - Chair of Psychiatry and Medical Psychology, Donetsk, Donetsk Oblast
  - Reg. Psychiatric Hospital, Odesa
  - Reg Cl.Ps.H.n.a.O.F. Malstev, Fem.Ac. Gen. Ps.D.5B, Poltava
  - CRI Cl.Psych.Hosp. #1, Fem. Psych. Dept. #2, Male I, Simferopol
  - Reg. Psych. Hosp.n.a.O.Yuschenko, Dept #21, Vinnitsia

REFERENCES:
- [Result] Loebel A, Cucchiaro J, Silva R, Kroger H, Hsu J, Sarma K, Sachs G. Lurasidone monotherapy in the treatment of bipolar I depression: a randomized, double-blind, placebo-controlled study. Am J Psychiatry. 2014 Feb;171(2):160-8. doi: 10.1176/appi.ajp.2013.13070984. PMID 24170180
- [Derived] Goldberg JF, Siu C, Tocco M, Pikalov A, Loebel A. The Effect of Lurasidone on Anxiety Symptoms in Patients With Bipolar Depression: A Post Hoc Analysis. J Clin Psychiatry. 2023 Jun 7;84(4):22m14732. doi: 10.4088/JCP.22m14732. PMID 37339360
- [Derived] Raison CL, Pikalov A, Siu C, Tsai J, Koblan K, Loebel A. C-reactive protein and response to lurasidone in patients with bipolar depression. Brain Behav Immun. 2018 Oct;73:717-724. doi: 10.1016/j.bbi.2018.08.009. Epub 2018 Aug 10. PMID 30102967
- [Derived] Sajatovic M, Forester BP, Tsai J, Kroger H, Pikalov A, Cucchiaro J, Loebel A. Efficacy of Lurasidone in Adults Aged 55 Years and Older With Bipolar Depression: Post Hoc Analysis of 2 Double-Blind, Placebo-Controlled Studies. J Clin Psychiatry. 2016 Oct;77(10):e1324-e1331. doi: 10.4088/JCP.15m10261. PMID 27529375
- [Derived] Rajagopalan K, Bacci ED, Ng-Mak D, Wyrwich K, Pikalov A, Loebel A. Effects on health-related quality of life in patients treated with lurasidone for bipolar depression: results from two placebo controlled bipolar depression trials. BMC Psychiatry. 2016 May 23;16:157. doi: 10.1186/s12888-016-0865-y. PMID 27215976
- [Derived] Chapel S, Chiu YY, Hsu J, Cucchiaro J, Loebel A. Lurasidone Dose Response in Bipolar Depression: A Population Dose-response Analysis. Clin Ther. 2016 Jan 1;38(1):4-15. doi: 10.1016/j.clinthera.2015.11.013. Epub 2015 Dec 22. PMID 26730454
- [Derived] Loebel A, Siu C, Rajagopalan K, Pikalov A, Cucchiaro J, Ketter TA. Recovery in bipolar depression: Post-hoc analysis of a placebo-controlled lurasidone trial followed by a long-term continuation study. J Affect Disord. 2015 Nov 1;186:376-82. doi: 10.1016/j.jad.2015.07.033. Epub 2015 Aug 5. PMID 26363720
- [Derived] McIntyre RS, Cucchiaro J, Pikalov A, Kroger H, Loebel A. Lurasidone in the treatment of bipolar depression with mixed (subsyndromal hypomanic) features: post hoc analysis of a randomized placebo-controlled trial. J Clin Psychiatry. 2015 Apr;76(4):398-405. doi: 10.4088/JCP.14m09410. PMID 25844756

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4/29/09 to 2/1/12
Groups:
- Placebo: Placebo : Placebo Comparator
- Lurasidone High Arm: lurasidone : lurasidone 20 mg/day for Days 1-2, 40 mg/day for Days 3-4, 60 mg/day for Days 5-6 and 80 mg/day on Day 7 and 80-120 mg/day
- Lurasidone Low Arm: lurasidone : lurasidone 20 mg/day for Days 1-7, beginning day 8 flexibly dosed 20-60 mg/day
Period: Overall Study
Arm/Group | Placebo | Lurasidone High Arm | Lurasidone Low Arm
Started | 170 | 169 | 166
Intent-to-Treat Population | 162 | 162 | 161
Safety Population | 168 | 167 | 164
Completed | 127 | 124 | 123
Not Completed | 43 | 45 | 43

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population is analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lurasidone High Arm | Lurasidone Low Arm | Total
Number analyzed (Participants) | 162 | 162 | 161 | 485
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 3 | 3
  Between 18 and 65 years | 159 | 159 | 155 | 473
  >=65 years | 3 | 3 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (12.45) | 42.0 (12.35) | 41.3 (12.31) | 41.5 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 98 | 91 | 276
  Male | 75 | 64 | 70 | 209
Region of Enrollment [Number; unit: participants]
  France | 5 | 4 | 4 | 13
  United States | 58 | 70 | 67 | 195
  Czech Republic | 19 | 19 | 17 | 55
  Ukraine | 16 | 17 | 16 | 49
  Romania | 9 | 2 | 4 | 15
  South Africa | 18 | 17 | 19 | 54
  Russian Federation | 10 | 10 | 11 | 31
  India | 27 | 23 | 23 | 73

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Endpoint (Week 6)
Description: Montgomery-Asberg Depression Rating Scale (MADRS)is a clinician-rated assessment of a subject's level of depression.
  The MADRS total score ranges from a minimum of 0 to a maximum of 60. For the MADRS total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome.
  The MADRS contains ten (10) items. The total score is computed as the sum of the scores for the 10 items.
Time Frame: Baseline to Week 6
Population: Intent-to-treat population is analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lurasidone High Arm | Lurasidone Low Arm
Number analyzed (Participants) | 162 | 162 | 161
units on a scale | -10.7 (0.83) | -15.4 (0.83) | -15.4 (0.83)
Statistical Analysis 1: Comparison: Placebo vs Lurasidone Low Arm; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -4.6, Standard Error of Mean 1.17 — A negative difference in least square mean change from baseline between Lurasidone group and placebo indicates a greater improvement in the Lurasidone group over the placebo group
Statistical Analysis 2: Comparison: Placebo vs Lurasidone High Arm; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -4.6, Standard Error of Mean 1.17 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Mean Change From Baseline to Endpoint (Week 6) in: Clinical Global Impression Bipolar Version, Severity of Illness (CGI-BP-S) Score (Depression)
Description: Clinical Global Impression Bipolar Version, Severity of Illness (CGI-BP-S) score (depression) is a clinician-rated assessment of a subject's level of depression.
  The CGI depression score ranges from a minimum of 0 to a maximum of 7. For the CGI depression score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome.
Time Frame: Baseline to Week 6
Population: Intent-to-treat population is analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lurasidone High Arm | Lurasidone Low Arm
Number analyzed (Participants) | 162 | 162 | 161
units on a scale | -1.14 (0.102) | -1.71 (0.101) | -1.83 (0.102)
Statistical Analysis 1: Comparison: Placebo vs Lurasidone Low Arm; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.69, Standard Error of Mean 0.143 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Lurasidone High Arm; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.57, Standard Error of Mean 0.143 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Change From Baseline to Endpoint (Week 6) in: Sheehan Disability Scale (SDS) Total Score
Description: Sheehan Disability Scale (SDS) total score is a subject-rated assessment of a subject's level of depression.
  The SDS total score ranges from a minimum of 0 to a maximum of 30. For the SDS total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome.
  The SDS contains three (3) items. The total score is computed as the sum of the scores for the 3 items.
Time Frame: Baseline to Week 6
Population: Intent-to-treat population is analyzed. Number of participants in table is not consistent with intent-to-treat population because: if one or more items are missing at a study visit, as can occur when a subject opts out of the work/school item because it does not apply, the authors of the scale recommend setting the total score to missing
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lurasidone High Arm | Lurasidone Low Arm
Number analyzed (Participants) | 100 | 105 | 88
units on a scale | -6.3 (0.77) | -9.8 (0.73) | -9.5 (0.81)
Statistical Analysis 1: Comparison: Placebo vs Lurasidone Low Arm; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Final Values) = -3.1, Standard Error of Mean 1.05 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Lurasidone High Arm; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -3.5, Standard Error of Mean 1.01 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: April 29,2009 - February 1, 2012
Description: Safety population is analyzed.
Arm/Group | Placebo | Lurasidone High Arm | Lurasidone Low Arm
Serious Adverse Events (participants affected / at risk) | 1/168 | 5/167 | 3/164
Other Adverse Events (participants affected / at risk) | 56/168 | 65/167 | 57/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=168) | Lurasidone High Arm (N=167) | Lurasidone Low Arm (N=164)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Panic Attack (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Restless Leg Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HIV Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous Absceses (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=168) | Lurasidone High Arm (N=167) | Lurasidone Low Arm (N=164)
Nausea (Gastrointestinal disorders) | 13 (87) | 29 (38) | 17 (24)
Headache (Nervous system disorders) | 20 (25) | 15 (16) | 23 (36)
Akathisia (Nervous system disorders) | 4 (6) | 18 (23) | 13 (18)
Insomnia (Psychiatric disorders) | 14 (19) | 11 (16) | 8 (12)
Somnolence (Nervous system disorders) | 7 (7) | 11 (13) | 7 (7)
Sedation (Nervous system disorders) | 3 (3) | 12 (13) | 5 (6)
Dizziness (Nervous system disorders) | 13 (13) | 10 (12) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.